CLINICAL TRIAL: NCT05605288
Title: Distal Versus Conventional Transradial Artery Access for Coronary Catheterization in Patients With ST-elevation Myocardial Infraction (STEMI): The DR-STEMI Trial
Brief Title: Distal Versus Conventional Transradial Artery Access for Coronary Catheterization in Patients With STEMI
Acronym: DR-STEMI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Patras (Other)
Responsible Party: Principal Investigator, Grigorios Tsigkas, Assistant Professor of Cardiology, University Hospital of Patras
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 26150/30.09.22
Record Dates: First submitted 2022-10-10; First posted 2022-11-04 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: ST Elevation Myocardial Infarction; Coronary Artery Disease; Distal Transradial Artery; Transradial Artery; Coronary Catheterization; Percutaneous Coronary Intervention; Primary PCI
Keywords: ST Elevation Myocardial Infarction; Coronary Artery Disease; distal transradial artery; transradial artery; coronary catheterization; percutaneous coronary intervention; primary PCI
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Coronary Artery Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Distal transradial artery access (Experimental): Vascular access after cannulation of distal transradial artery through anatomical snuffbox for coronary angiography and interventions
  Interventions: Procedure: Coronary angiography +/- percutaneous coronary intervention
- Conventional transradial artery access (Active Comparator): Vascular access after puncturing on the conventional transradial artery for performing coronary angiography and interventions
  Interventions: Procedure: Coronary angiography +/- percutaneous coronary intervention

INTERVENTIONS:
Procedure: Coronary angiography +/- percutaneous coronary intervention — Coronary angiography +/- percutaneous coronary intervention

SUMMARY:
Recently, a novel distal transradial, through anatomical snuffbox, approach has been proposed for undertaking percutaneous coronary angiography and interventions. The existing literature has evaluated distal transradial access (dTRA) as a feasible and safe approach, with faster hemostasis, lower rates of periprocedural complications and reduced incidence of radial artery occlusion (RAO). Aim of the present study is to compare dTRA versus conventional TRA access in patients with STEMI undergoing coronary angiography and interventions regarding peri- and post-procedural characteristics.

DETAILED DESCRIPTION:
Gaining vascular access is the first, mandatory step for undertaking percutaneous coronary angiography and interventions. The recent guidelines, published by European Society of Cardiology (ESC), American College of Cardiology (ACC), American Heart Association (AHA) and Society for Cardiovascular Angiography and Interventions (SCAI), propose TRA as the gold standard for acute coronary syndromes (ACS), chronic coronary syndrome (CCS) percutaneous coronary interventions (PCI). Recently, a novel distal transradial, through anatomical snuffbox, approach has been proposed. The existing literature has evaluated distal transradial access (dTRA) as a feasible and safe approach, with faster hemostasis, lower rates of periprocedural complications and reduced incidence of radial artery occlusion (RAO). Mutual point of all the previous RCTs is that excluded patients suffering from ST-elevation Myocardial Infraction (STEMI). Aim of the present study is to compare dTRA versus conventional TRA access in patients with STEMI undergoing coronary angiography and interventions regarding peri- and post-procedural characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Indication: ST-Elevation Myocardial Infraction

Exclusion Criteria:

* Non-palpable radial artery
* Previous CABG
* Anatomical restrictions for forearm approach
* Hemodynamic instability
* Previous radial artery catheterization from the same arm during the last 30-days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 554 (Estimated)
Dates: Start 2024-05-23 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
needle-to-wire time | Immediately post-procedurally
  needle-to-wire time

SECONDARY OUTCOMES:
Radial artery occlusion using Doppler examination prior to hospital discharge | The evaluation will be performed during hospitalization for STEMI and prior discharge, typically the 4th day after PCI
  Radial artery patency evaluation with Doppler ultrasound prior to hospital discharge for detecting possible occlusion after cannulation
Access site crossover rate | Immediately post-procedurally
  Crossover rate from distal transradial artery access to other access point
Sheath insertion time | Immediately post-procedurally
  Duration required from the beginning of puncture until sheath insertion
Total procedure time | Immediately post-procedurally
  Total duration of coronary angiography and angioplasty
The time interval between the initiation of radial artery puncture and the completion of coronary angiography, until the beginning of the possible PCI | Immediately post-procedurally
  The time interval between the initiation of radial artery puncture and the completion of coronary angiography, until the beginning of the possible PCI
Required time for coronary angiography completion, after sheath insertion | Immediately post-procedurally
  Required time for coronary angiography completion, after sheath insertion
Required time percutaneous coronary intervention completion | Immediately post-procedurally
  Required time percutaneous coronary intervention completion
Total fluoroscopy time | Immediately post-procedurally
  Total fluoroscopy time
Total Dose Area Product (DAP) | Immediately post-procedurally
  Total Dose Area Product (DAP)
Air Kerma | Immediately post-procedurally
  Air Kerma
Hemostasis time | 3 hours
  Time required for achieving hemostasis
Vascular complications | 24 hours
  Vascular complications
Hematomas classification (modified EASY classification) | 24 hours
  Hematomas classification using modified EASY which is compatible with dTRA
30-days Clinical follow-up (on site or via telephone call) | 30 days
  30-days Clinical follow-up (on site or via telephone call)

CONTACTS AND LOCATIONS:
Overall Officials: Grigorios Tsigkas, MD, PhD, Principal Investigator — University Hospital of Patras; Adel Aminian, MD, PhD, Principal Investigator — Centre Hospitalier Universitaire de Charleroi; Juan Inglesias, MD, PhD, Principal Investigator — Department of Cardiology, Geneva University Hospitals, Geneva, Switzerland.
Locations (3):
- Department of Cardiology, Centre Hospitalier Universitaire de Charleroi, Charleroi, Belgium
- University Hospital of Patras, Pátrai, Greece
- Department of Cardiology, Geneva University Hospitals, Geneva, Switzerland., Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tsigkas G, Moulias A, Papageorgiou A, Ntouvas I, Grapsas N, Despotopoulos S, Apostolos A, Papanikolaou A, Smaili K, Vasilagkos G, Davlouros P, Hahalis G. Transradial access through the anatomical snuffbox: Results of a feasibility study. Hellenic J Cardiol. 2021 May-Jun;62(3):201-205. doi: 10.1016/j.hjc.2020.02.002. Epub 2020 Mar 2. PMID 32135274
- [Background] Didagelos M, McEntegart M, Kouparanis A, Tsigkas G, Koutouzis M, Tsiafoutis I, Kassimis G, Oldroyd KG, Ziakas A. Distal Transradial (Snuffbox) Access for Coronary Catheterization: A Systematic Review. Cardiol Rev. 2021 Jul-Aug 01;29(4):210-216. doi: 10.1097/CRD.0000000000000339. PMID 34061817
- [Background] Sgueglia GA, Hassan A, Harb S, Ford TJ, Koliastasis L, Milkas A, Zappi DM, Navarro Lecaro A, Ionescu E, Rankin S, Said CF, Kuiper B, Kiemeneij F. International Hand Function Study Following Distal Radial Access: The RATATOUILLE Study. JACC Cardiovasc Interv. 2022 Jun 27;15(12):1205-1215. doi: 10.1016/j.jcin.2022.04.023. Epub 2022 May 17. PMID 35595672
- [Background] Eid-Lidt G, Rivera Rodriguez A, Jimenez Castellanos J, Farjat Pasos JI, Estrada Lopez KE, Gaspar J. Distal Radial Artery Approach to Prevent Radial Artery Occlusion Trial. JACC Cardiovasc Interv. 2021 Feb 22;14(4):378-385. doi: 10.1016/j.jcin.2020.10.013. PMID 33602433
- [Background] Tsigkas G, Papageorgiou A, Moulias A, Kalogeropoulos AP, Papageorgopoulou C, Apostolos A, Papanikolaou A, Vasilagkos G, Davlouros P. Distal or Traditional Transradial Access Site for Coronary Procedures: A Single-Center, Randomized Study. JACC Cardiovasc Interv. 2022 Jan 10;15(1):22-32. doi: 10.1016/j.jcin.2021.09.037. Epub 2021 Dec 15. PMID 34922888
- [Background] Tsigkas G, Papageorgiou A, Moulias A, Apostolos A, Kalogeropoulos AP, Davlouros P. Reply: Distal Transradial Access for Primary PCI in ST-Segment Elevation Myocardial Infarction. JACC Cardiovasc Interv. 2022 Apr 11;15(7):795-796. doi: 10.1016/j.jcin.2022.02.039. No abstract available. PMID 35393114
- [Background] Aminian A, Sgueglia GA, Wiemer M, Kefer J, Gasparini GL, Ruzsa Z, van Leeuwen MAH, Ungureanu C, Leibundgut G, Vandeloo B, Kedev S, Bernat I, Ratib K, Iglesias JF, Al Hage E, Posteraro GA, Pascut D, Maes F, Regazzoli D, Kakonyi K, Meijers TA, Colletti G, Krivoshei L, Lochy S, Zafirovska B, Horak D, Nolan J, Degrauwe S, Tobita K, Saito S. Distal Versus Conventional Radial Access for Coronary Angiography and Intervention: The DISCO RADIAL Trial. JACC Cardiovasc Interv. 2022 Jun 27;15(12):1191-1201. doi: 10.1016/j.jcin.2022.04.032. Epub 2022 May 17. PMID 35595673
- [Background] Tsigkas G, Apostolos A, Davlouros P. Less Is More, But Not Always: Distal Transradial Access for Radial Artery Occlusion Prevention. JACC Cardiovasc Interv. 2022 Jun 27;15(12):1202-1204. doi: 10.1016/j.jcin.2022.05.001. Epub 2022 May 17. No abstract available. PMID 35583362
- [Derived] Tsigkas G, Trigka-Vasilakopoulou A, Apostolos A, Papafaklis M, Colletti G, Mugnolo A, Ruzsa Z, Ungureanu C, Nikas D, Xaplanteris P, Gasparini GL, Sciahbasi A, Tsiafoutis I, Poulimenos LE, Didagelos M, Pappas L, Stougiannos P, Hamilos M, Ziakas A, Timpilis F, Karanasos A, Moulias A, Sgueglia GA, Aminian A, Iglesias JF, Michalis L, Davlouros P. Distal versus conventional transradial artery access for coronary catheterization in patients with STEMI (DR-STEMI): Rationale and design of an international, multicenter, randomized trial. Am Heart J. 2026 Jan;291:73-80. doi: 10.1016/j.ahj.2025.08.007. Epub 2025 Aug 13. PMID 40816555